CLINICAL TRIAL: NCT03763201
Title: Role of Glucocorticoid-induced Tumour Necrosis Factor Receptor Related Protein (GITR) as a Marker of Activity in Rheumatoid Arthritis Patients
Brief Title: Glucocorticoid-induced Tumour Necrosis Factor Receptor Related Protein (GITR) in Rheumatoid Arthritis
Acronym: GITR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Other Study IDs: BenhaU 112018
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; glucocorticoid-induced tumour necrosis factor receptor related protein
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and synovial fluid samples from RA patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatoid arthritis: recently diagnosed rheumatoid arthritis patients in whom we measure Glucocorticoid-induced Tumour Necrosis Factor Receptor Related Protein (GITR) in their serum and synovial fluid (if clinically determined knee effusion)
  Interventions: Diagnostic Test: measurement of GITR
- control group: age and sex matched healthy volunteers whom we measure Glucocorticoid-induced Tumour Necrosis Factor Receptor Related Protein (GITR) in their serum.
  Interventions: Diagnostic Test: measurement of GITR

INTERVENTIONS:
Diagnostic Test: measurement of GITR — serum and synovial fluid measurement of glucocorticoid-induced tumour necrosis factor receptor related protein

SUMMARY:
This study aimed to measure serum and synovial fluid (SF) levels of GITR in patients with recent onset RA before and after initiation of therapy

DETAILED DESCRIPTION:
1. Technical design:

   Study design: a longitudinal observational cohort study.

   This study will be carried out on two groups:
   * Group (I): fifty early onset rheumatoid arthritis (RA) patients fulfilled the 2010 American college of rheumatology (ACR) - European league against rheumatism (EULAR) classification criteria for RA [11].
   * Group (II): Twenty healthy individuals of matching age and sex as control group.

   Both groups will be recruited from the in-patients and out-patients' clinic of the Rheumatology, Rehabilitation& Physical Medicine Department, Benha University Hospital.

   All patients will be evaluated at baseline at 6 months follow up using:

   (A) Clinical evaluation 1. Complete history taking. 2. Thorough clinical examination. 3. Disease activity using DAS28 [12]

   (B) Laboratory assessment:

   All patients will be subjected to the following measurements:
   1. Erythrocyte sedimentation rate (ESR).
   2. C reactive protein (CRP).
   3. Rheumatoid factor (RF)
   4. Anti-cyclic citrullinated peptide (Anti- CCP).
   5. glucocorticoid-induced tumour necrosis factor receptor related protein (GITR)

   (D) Musculoskeletal ultrasound assessment: Ultrasound examinations will be performed for patients and control groups using a Logiq e equipped with a broadband 8- to 13-MHz linear transducer
2. Statistical analysis The collected data will be tabulated and analyzed using suitable statistical computer version.

ELIGIBILITY:
Inclusion Criteria:

* fulfill 2010 criteria for classification of rheumatoid arthritis recentely diagnosed

Exclusion Criteria:

* infection malignancy receiving treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 2 groups: first: recently diagnosed RA patients 2nd : healthy control ( age and sex matched)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
28 tender joints count | 4 months
  tender joints count of both shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees in Rheumatoid patients
28 swollen joints count | 4 months
  swollen joints count of both shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees in Rheumatoid patients
patient's global assessment of disease activity | 4 months
  patient's global assessment of disease activity on 0 to 100 mm VAS 0 is the best and 100 is the worst.
disease activity score of 28 joint count (DAS28) | 4 months
  DAS28 is calculated from tender and swollen joint counts , ESR and patient's global assessment of disease activity according to the following formula DAS28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * global patient assesment
erythrocyte sedimentation rate (ESR) | 4 months
  ESR measured in mm/1st hour by westergren method
C reactive protein (CRP) | 4 months
  CRP measured in mg/L using nephlometry
grey scale12 joint score | 4 months
  grey scale musculoskeletal ultrasound including bilateral examination of both 2nd metacarpophalengeal (MCP) joints, 3rd MCP joints, wrists, elbows, knees and ankles then the following greyscale synovitis semiquantitative grades were assumed: Grade 0: absent. Grade 1: mild with anechoic / hypoechoic line below the capsule of the joint. Grade 2: moderate with elevation of the joint capsule that becomes parallel to the area of the joint. Grade 3: severe with marked distension of the capsule.
power Doppler 12 joint score | 4 months
  power Doppler musculoskeletal ultrasound including bilateral examination of both 2nd metacarpophalengeal (MCP) joints, 3rd MCP joints, wrists, elbows, knees and ankles then the following power Doppler synovitis grades were assumed: Grade 0: no colour signal inside joint area. Grade 1: up to 3 colour signals inside joint area. Grade 2: colour signals less than half of joint area and more than grade 1. Grade 3: colour signals more than half of joint area.
rheumatoid factor | 4 months
  rheumatoid factor measured in U/ml using latex agglutination test
anticyclic citrullinated antibody (Anti CCP) | 4 months
  Anti CCP measured in Unit/ml using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Waleed A Hassan, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- bENHA UNIVERSITY HOSPITAL, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided